CLINICAL TRIAL: NCT06162676
Title: Pilot Testing of a Game-Based Intervention to Promote HPV Vaccination in Families With Unvaccinated Children
Brief Title: Game-Based Intervention to Promote HPV Vaccination
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: Arizona State University (Other)
Responsible Party: Principal Investigator, Angela Chia-Chen Chen, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: STUDY00009385
Record Dates: First submitted 2023-11-30; First posted 2023-12-08 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: HPV Infection; Vaccine-Preventable Diseases
Keywords: adolescent, parent, game intervention, HPV prevention
MeSH Terms: conditions — Papillomavirus Infections; Vaccine-Preventable Diseases

STUDY DESIGN:
Intervention Model Description: intervention vs. usual care (control)
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HPV game group (Experimental): Parent-child dyads receive a HPV game intervention
  Interventions: Behavioral: HPV game
- Usual care (No Intervention): Parent-child dyads receive child's usual care

INTERVENTIONS:
Behavioral: HPV game — A brief health game for parent-child dyads to promote child's HPV vaccination
  Arms: HPV game group

SUMMARY:
This study will examine the feasibility and acceptability of an innovative game-based intervention designed for families of youth aged 11-14 to promote HPV vaccination; will explore changes in key outcomes and related measures; and will identify factors contributing to or impeding effective implementation in health clinic settings. The intervention and its approach have the potential to reduce health disparities in HPV-associated cancers in youth via low-cost technology and timely intervention.

DETAILED DESCRIPTION:
Guided by Social Cognitive Theory, we propose to

1. examine the feasibility and acceptability of a new HPV preventive intervention, the HPV Detective video game, designed for youth and their parents;
2. explore pre-post, intervention-related change in vaccine intent and uptake as well as change in theoretically posited intervention mediators; and
3. assess the potential for broader intervention implementation. Using a sequential mixed-methods, 2-group (intervention vs usual care), longitudinal design, 64 parent-youth dyads (32/per study condition) will be recruited.

Parent-youth dyads in the intervention will play HPV Detective (tablet format) at the clinic prior to the healthcare provider visits. The control dyads will receive standard clinic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Youth: (1) 11-14 years old; (2) have not received the 1st dose of HPV vaccine; (3) speak and read English
* Parent: (1) are the parent/legal guardian of the participating child; (2) ≥ 18 years old; (3) speak English or Spanish; (4) own a smartphone; (5) agree to participate in the research activities at study sites; (6) agree to receive text messages.
* Healthcare providers: (1) ≥ 20 years old; (2) speak English or Spanish); (3) work at study sites

Exclusion Criteria:

* Individuals are unable to comprehend the consent or assent forms due to cognitive issues

Ages: 11 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 131 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-07-30 (Actual); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Percentage of eligible individuals agreeing to participate | 2 years
  Assessed by the % of eligible individuals agreeing to participate
Percentage of eligible individuals who complete the intervention (intervention arm only) and assessments (all participants) | 2 years
  Assessed by the % of eligible individuals who complete the intervention and assessments
Ease of use (intervention arm only) | 2 years
  (1) device-recorded time to complete interactive modules and the full game; (2) self reported easy of use
Parent and child acceptability of the intervention (intervention arm only) | 2 years
  Assessed by a 12-item Likert scale.
Intention to vaccinate the child against HPV | 2 years
  Assessed by a Likert scale question: how likely will you (parent) vaccinate your child against HPV? Responses: (1) Very unlikely to (5) Very likely
Child vaccination status (1st & 2nd doses). | 2 years
  Assessed by one binary (yes/no) question regarding whether or not the child has received the 1st & 2nd dose of HPV vaccine.

CONTACTS AND LOCATIONS:
Overall Officials: ANGELA CHEN, PhD, Principal Investigator — Michigan State University
Locations (1):
- Michigan State University, East Lansing, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
This study will provide de-identified survey data stored in an encrypted electronic database. They will be available free of identifiers to avoid the possibility of disclosing identify of research participants. Quantitative data collected from this study will be made available to qualified scientists for research purposes following acceptance for publication of the main findings derived from the final data set.
Supporting Information: SAP
Time Frame: The data will be available when the award ends and following acceptance for publication of the main findings derived from the final data set. It will be available for 10 years.
Access Criteria: The data will remain the property of the provider; the recipient shall show proof of appropriate training in the responsible conduct of research; any publication resulting from use of the data will acknowledge the provider and NIH of the original project from which the data were derived; the data will not be used for commercial or for-profit purposes; the data will not be further distributed to others; the provider makes no representations and extends no warranties of any kind, either expressed or implied; the recipient shall assume all liability for claims for damages against it by third parties that may arise from the use of the data; the recipient agrees to pay the cost of preparation and distribution of the data. Availability and use of the data may be limited by additional local institutional review board policies or by local, state, and federal laws and regulations.